CLINICAL TRIAL: NCT03852953
Title: Under- and Overdiagnosis in BreastScreen Norway
Status: Completed | Type: Observational
Sponsor: Norwegian Institute of Public Health (Other Government)
Collaborators: Extrastiftelsen (Other)
Responsible Party: Sponsor
Other Study IDs: 17/222; 2018/FO201362 (Other Grant/Funding Number: ExtraStiftelsen)
Record Dates: First submitted 2018-11-12; First posted 2019-02-25 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2021-01

CONDITIONS: Breast Cancer
Keywords: Screening; Mammography; Overdiagnosis; Womens' perspectives; Harms and benefits; False negative; Quantitative methods; Survival
MeSH Terms: conditions — Breast Neoplasms | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Study 1: Under- and overdiagnosed group: Non-proportional stratified sample of women diagnosed with interval or screen-detected breast cancers after participation in BreastScreen Norway. This sample will include under- or overdiagnosed cancers, as well as cancers that were not under- or overdiagnosed.
  Interventions: Other: Under- or overdiagnosed cancer
- Study 2: Rate of overdiagnosis group: Women residing in Norway, born between 1927 and 1934 (inclusive). This cohort will include women who have attended screening and who have not attended screening.
  Interventions: Other: Screening
- Study 3: Awareness and knowledge group: Women aged 50-69, and practising family doctors aged 25-75, currently living in Norway.

INTERVENTIONS:
Other: Under- or overdiagnosed cancer — Diagnosed with a cancer that was visible on prior mammograms
  Groups: Study 1: Under- and overdiagnosed group
Other: Screening — Invited or attended BreastScreen Norway
  Groups: Study 2: Rate of overdiagnosis group

SUMMARY:
This PhD project will describe tumour characteristics and survival associated with of under- and overdiagnosed breast cancers, the rate of overdiagnosis in BreastScreen Norway, and whether women and family doctors are aware of, and knowledgeable about, under- and overdiagnosis in breast cancer screening.

DETAILED DESCRIPTION:
Mammographic screening among women aged 50-69 reduces breast cancer mortality but also carries some risk. This PhD project will study under- and overdiagnosis, two risks associated with mammographic screening, in BreastScreen Norway. Underdiagnosis can occur when a tumour is present but not detected as a result of screening, while overdiagnosis can occur when a woman is diagnosed with a slow growing cancer that would not become symptomatic during her lifetime.

This project will address the following topics and research questions using observational study methods.

Study 1: To determine whether tumour histopathology and survival differentially associated with potentially under- or overdiagnosed interval and screen-detected breast cancers.

* Do women with potentially underdiagnosed interval cancers have different tumour histopathology and survival than those whose interval cancers showed no signs at the prior screen?
* Do women with potentially overdiagnosed screen-detected cancer have different tumour histopathology and survival than those whose screen-detected cancer showed no signs at the prior screen?

Study 2: To estimate overdiagnosis in the screening program using individual-level data:

* What was the rate of overdiagnosis for women screened in the program during 1996-2003?
* How does adjusting for sociodemographic factors affect estimates of overdiagnosis?

Study 3: To describe awareness and knowledge about under- and overdiagnosis and breast screening in general:

* Are women aware of and knowledgeable about under- and overdiagnosis in breast screening?
* Are family doctors aware of and knowledgeable about breast screening, and under- and overdiagnosis? Are they confident in their ability to relay this information to their patients?

Study 1 is a quality improvement study and has approval from Personvernombudet (PVO 2016-4696). Study 2 has research ethics board (REK) approval (REK 2013/795), while REK approval will be sought for Study 3.

ELIGIBILITY:
Study 1

Inclusion Criteria:

* Breast cancer diagnosed within BreastScreen Norway using digital mammography
* Prior screening images available for review

Study 2

Inclusion Criteria:

* Women born between 1927 and 1934 (inclusive)
* Legal resident in Norway at any time between 1996 and 2003 (inclusive)

Study 3

Inclusion Criteria:

* Women residing in Norway, aged 50-69 (inclusive)
* Practising family doctors in Norway, aged 25-75 (inclusive)
* Provide informed consent

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women aged 50-69, and practising female and male family doctors aged 25-75, residing in Norway.
Sampling Method: Non-Probability Sample
Enrollment: 3915 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-06-08 (Actual); Study Completion 2020-06-08 (Actual)

PRIMARY OUTCOMES:
Study 1: Prognostic and predictive histopathologic characteristics | At time of diagnosis
  - Histopathological type (Ductal carcinoma in situ, invasive carcinoma of no special type, invasive lobular carcinoma)
Study 1: Prognostic and predictive histopathologic characteristics | At time of diagnosis
  - Maximum tumour diameter (mm)
Study 1: Prognostic and predictive histopathologic characteristics | At time of diagnosis
  - Tumour grade (1, 2, 3)
Study 1: Prognostic and predictive histopathologic characteristics | At time of diagnosis
  - Lymph node involvement (Yes/No)
Study 1: Prognostic and predictive histopathologic characteristics | At time of diagnosis
  - Receptor status (Positive/Negative)
Study 1: Prognostic and predictive histopathologic characteristics | At time of diagnosis
  - Ki67 expression (0-100%)
Study 2: Crude and adjusted rate of overdiagnosis | 1996 to 2016
  - Crude and adjusted measures of overdiagnosis will be presented to show the amount and direction of confounding resulting from sociodemographic factors.
Study 3: Agreement between awareness and knowledge of overdiagnosis | One day (Measurements taken once at time of survey completion)
  Agreement between awareness (yes versus no/incomplete) and knowledge (yes versus no/incomplete) of overdiagnosis

SECONDARY OUTCOMES:
Study 1: Survival | Date of diagnosis until 31 December 2017
  - Overall survival
Study 1: Survival | Date of diagnosis until 31 December 2017
  - Breast cancer specific survival

OTHER OUTCOMES:
Study 3: Factors associated with awareness and knowledge of overdiagnosis | One day (Measurements taken once at time of survey completion)
  Using a self-administered web-based questionnaire designed for this study, the investigators will analyse survey responses to determine whether self-reported age (categorised into 5-year age groups) is associated with awareness and knowledge of overdiagnosis. This will be done separately for women and family doctors.
Study 3: Factors associated with awareness and knowledge of overdiagnosis | One day (Measurements taken once at time of survey completion)
  Using a self-administered web-based questionnaire designed for this study, the investigators will analyse survey responses to determine whether self-reported formal education (none; primary school; high school; up to 4 years postsecondary; more than 4 years of postsecondary education) is associated with awareness and knowledge of overdiagnosis among women.

CONTACTS AND LOCATIONS:
Overall Officials: Solveig Hofvind, PhD, Principal Investigator — Norwegian Institute of Public Health
Locations (1):
- Cancer Registry of Norway, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hovda T, Tsuruda K, Hoff SR, Sahlberg KK, Hofvind S. Radiological review of prior screening mammograms of screen-detected breast cancer. Eur Radiol. 2021 Apr;31(4):2568-2579. doi: 10.1007/s00330-020-07130-y. Epub 2020 Oct 1. PMID 33001307
- [Result] Tsuruda KM, Hovda T, Bhargava S, Veierod MB, Hofvind S. Survival among women diagnosed with screen-detected or interval breast cancer classified as true, minimal signs, or missed through an informed radiological review. Eur Radiol. 2021 May;31(5):2677-2686. doi: 10.1007/s00330-020-07340-4. Epub 2020 Nov 12. PMID 33180162
- [Result] Tsuruda KM. Overdiagnosis and 'underdiagnosis' in BreastScreen Norway [dissertation]. [Oslo, Norway]: University of Oslo; 2021. 108 p. Available at: http://urn.nb.no/URN:NBN:no-91337
- See also: Project description on Extrastiftelsen's website (Norwegian) — https://www.extrastiftelsen.no/prosjekter/over-og-underdiagnostisering-i-mp/
- See also: Project description on the Cancer Registry of Norway's website (English/Norwegian) — https://www.kreftregisteret.no/en/Research/Projects/over--og-underdiagnosis-in-breastscreen-norway/
- See also: Article about study with interview (Norwegian; pages 23-24) — https://www.brystkreftforeningen.no/getfile.php/134688-1615383992/Athene/Athene-2018-01.pdf